CLINICAL TRIAL: NCT06247319
Title: A Non-interventional, Prospective Study to Evaluate the Effectiveness of Risankizumab in Patients With Recent Diagnosis of Moderate Plaque Psoriasis in a Real Life Setting in Greece- the REDEFINE Study
Brief Title: Study to Evaluate the Effectiveness of Risankizumab in Participants With a Recent Diagnosis of Moderate Plaque Psoriasis in a Real-life Setting in Greece
Acronym: REDEFINE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-179
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Moderate Plaque Psoriasis; Moderate Psoriasis; Psoriasis
Keywords: Moderate Psoriasis; Psoriasis; Moderate Plaque Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated with Risankizumab: Participants with a recent diagnosis of moderate plaque PsO (defined as ≤24 months since the first diagnosis of moderate PsO), and naïve to advanced treatments (biologics, apremilast, and deucravacitinib) will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
Psoriasis is a skin disorder wherein skin cells multiply faster than normal, making the skin itchy and look patchy and red. It is caused by an overactive immune system where the body attacks healthy tissue by mistake. The impact of Psoriasis on quality of life can be significant, especially in moderate-to-severe disease which affects approximately half of the participants with plaque Psoriasis. Participants with Psoriasis are marked by their disease physically, psychologically, and emotionally. In addition to the above, their disease exerts a negative effect on various dimensions of health-related quality of life such as daily activities and work productivity. This study is designed to provide information regarding the impact of risankizumab on short-term and long-term clinical parameters of Psoriasis as well as the patient-reported outcomes (PROs) in participants with a recent diagnosis (less than or equal to 24 months) of moderate Psoriasis who are naïve to advanced treatments.

Risankizumab is an approved drug for the treatment of Plaque Psoriasis. Approximately 250 participants with a recent diagnosis of moderate plaque psoriasis (defined as less than or equal to 24 months since the first diagnosis of moderate Psoriasis), and naïve to advanced treatments (biologics, apremilast, and deucravacitinib) will be enrolled at approximately 20 sites in Greece.

Participants will receive risankizumab as prescribed by their treating dermatologist in accordance with local authorization and independently from the study. Participants will be enrolled and observed for approximately two years.

There is expected to be no additional burden for participants in this trial. Study visits comprised of private practices and hospital clinics as per standard of care.

DETAILED DESCRIPTION:
Any of a variety of other sampling processes, such as convenience sampling or invitation to volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed diagnosis of moderate plaque PsO made by a specialist ≤24 months prior to risankizumab prescription defined as:

  * Percentage of body surface affected by PsO Body Surface Area (BSA) >2% and <20%
  * Psoriasis Area and Severity Index (PASI) score >10
  * Static Physician's Global Assessment (sPGA) score =3 (moderate) based on a 5-point scale (0-4)
* Participants naïve to advanced treatments (biologics, apremilast, and deucravacitinib)
* Participants who have been prescribed treatment with risankizumab in line with marketing authorization and local access conditions, prior to signed Informed Consent
* Decision to treat with risankizumab has been made independently and prior to enrolment in the study
* Participants must be willing and able to read and complete the study specific questionnaires

Exclusion Criteria:

* Participants who currently receive treatment with any investigational drug/device/intervention or who have received any investigational product within 30 days before risankizumab initiation
* Pregnancy or lactation
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a recent diagnosis of moderate plaque PsO (defined as ≤24 months since the first diagnosis of moderate PsO), and naïve to advanced treatments (biologics, apremilast, and deucravacitinib) treated with Risakizumab according to local label.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Psoriasis Area and Severity Index (PASI) score less than or equal to 2 | Baseline to Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
Proportion of participants achieving a Dermatology Life Quality Index (DLQI) score of 0 or 1 (include only patients with DLQI score less than or equal to 2 at Baseline) | Baseline to Week 16
  DLQI (Dermatology Life Quality Index) assesses symptoms and impacts of dermatologic diseases on quality of life. DLQI scores range from 0 (no effect) to 30 (very large effect), with a higher score indicating a more impaired quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (22):
- Greece (22):
  - Olympion General Clinic /ID# 266258, Pátrai, Achaia
  - Iatriko Psichikou /ID# 272851, Athens, Attica
  - 251 Hellenic Air Force General Hospital /ID# 268135, Athens, Attica
  - University General Hospital Attikon /ID# 263442, Athens, Attica
  - General Hospital Andreas Syggros /ID# 263443, Athens, Attica
  - General Hospital Andreas Syggros /ID# 266248, Athens, Attica
  - Tzaneio Prefecture General Hospital of Piraeus /ID# 263448, Piraeus, Attica
  - Asklipieio General Hospital of Voula /ID# 268136, Voula, Attica
  - University General Hospital of Heraklion /ID# 268777, Heraklion, Crete
  - Venizelio Regional General Hospital of Heraklion /ID# 268778, Heraklion, Irakleio
  - Konstantopoulio General Hospital /ID# 266257, Nea Ionia, Magnisia
  - West Attica General Hospital "Agia Varvara" /ID# 266256, Agía Varvára
  - 401 General Military Hospital /ID# 277393, Athens
  - Hygeia Hospital /ID# 263455, Athens
  - KAT Attica General Hospital /ID# 266249, Kifissia
  - University General Hospital of Larissa /ID# 263440, Larissa
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 262530, Thessaloniki
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 263452, Thessaloniki
  - General Hospital of Thessaloniki "Agios Pavlos'' /ID# 267506, Thessaloniki
  - Papageorgiou General Hospital /ID# 262529, Thessaloniki
  - General Hospital of Tripoli Panarkadiko "Evangelistria" /ID# 266251, Tripoli
  - General Hospital of Xanthi /ID# 268133, Xánthi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-179